CLINICAL TRIAL: NCT00525226
Title: Perinatal Stress and Gene Influences: Pathways to Infant Vulnerability
Brief Title: Evaluating the Effects of Stress in Pregnancy
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael J. Owens, Professor, Psychiatry, Emory University
Other Study IDs: IRB00004249; P50MH077928 (NIH); DDTR B3-PDB
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Depression; Panic Disorder; Generalized Anxiety Disorder; Post-Traumatic Stress Disorder; Obsessive Compulsive Disorder (OCD)
Keywords: Psychiatry; Psychology; Pregnancy; Stress; Anxiety
MeSH Terms: conditions — Depression; Panic Disorder; Generalized Anxiety Disorder; Stress Disorders, Post-Traumatic; Obsessive-Compulsive Disorder; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasm, serum, and urine samples are processed and stored at each research visit.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Women who have experienced symptoms of depression or anxiety during pregnancy.

SUMMARY:
This study will evaluate pregnant women with a past or current diagnosis of depression or anxiety to gain a better understanding of how these disorders can affect an infant's development, both during and after pregnancy.

DETAILED DESCRIPTION:
Depression and anxiety are serious conditions affecting millions of people each year. In fact, it is estimated that approximately one in every four women will be treated for a mood disorder, such as depression or anxiety, at some point in her life. As effective treatment options continue to develop, many women diagnosed with depression or anxiety are able to resume normal lives and may choose to become pregnant. However, studies suggest that the intrauterine environment can be altered by maternal stress, depression, and anxiety, which may affect the fetus during pregnancy. Also, antidepressant medications have been known to cause complications for both the mother and fetus, which can make pregnancy a very difficult time for women with a history of depression and anxiety. These women are more prone to relapse during pregnancy, even if they previously recovered from the disorder. The purpose of this study is to evaluate whether symptoms of depression and anxiety, during or soon after pregnancy, affect an infant's social and emotional development.

Participation in this study will occur from early in the woman's pregnancy until her infant's first birthday. Participants will attend at least eight study visits during pregnancy and five study visits during the first year of the infant's life. Most study visits will take place at the Emory University clinic on campus. During the first study visit, participants will complete questionnaires regarding their current mood, stressors, supports, experiences during pregnancy, symptoms of depression or anxiety, and any treatment or medications they are currently receiving. Urine and blood will also be collected at the initial visit. Follow-up visits, lasting 1 hour, will occur monthly until delivery. During these visits, similar questionnaires will be administered and blood, urine, and saliva samples will be collected. Uterine blood flow, fetal activity, and fetal heart rate will be recorded at some follow-up visits. Women who undergo an amniocentesis will have the option of providing a sample of amniotic fluid and an additional blood sample.

Immediately after delivery, blood from the baby's umbilical cord and blood from the mother will be collected. A week after delivery, a home visit will be scheduled to assess each mother's mood, stress, supports, delivery complications, and first impressions of the new baby. At this time, a behavioral assessment will also be conducted on each infant, and mothers will be observed while interacting with their child. At the infant's 6-month pediatrician visit, a saliva sample will be taken to measure levels of cortisol and other indicators of stress. Infants will be assessed at three other times before their first birthday. During these assessments, the infant's ability to regulate his or her emotions will be evaluated by videotaped behavioral observations, stress hormones from saliva, heart rate, or recordings of brain activity through the use of either an electroencephalogram (EEG) or event related potentials (ERP). Lastly, participants will be given the option to provide a DNA sample for further analysis and future research. Fathers of the babies will be included in selected study visits. Results from this study will be used to help prevent emotional and social developmental problems in infants whose mothers have been diagnosed with either depression or anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for major depressive disorder, panic disorder, obsessive-compulsive disorder, generalized anxiety disorder, or post-traumatic stress disorder
* Planning pregnancy or less than 16 weeks pregnant by last menstrual period
* Written and verbal fluency in English
* Known identity of biological father

Exclusion Criteria:

* Suicidal or homicidal
* Psychosis
* Meets DSM-IV criteria for bipolar disorder, schizophrenia, or an eating disorder
* Alcohol or substance abuse within 6 months prior to study start date
* Current illness requiring treatment that can influence outcomes (e.g., epilepsy, asthma, autoimmune disorders)
* Abnormal thyroid stimulating hormone
* Anemic

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of child bearing potential between the ages of 18 to 45 years of age with or without a history of depression or anxiety disorders.
Sampling Method: Non-Probability Sample
Enrollment: 1431 (Actual)
Dates: Start 2007-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Social and emotional development of infants who have mothers with depression and anxiety, during or soon after pregnancy | Measured at Year 1 post-pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Zachary N. Stowe, MD, Principal Investigator — Emory University; Michael J Owens, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Women's Mental Health Program, Atlanta, Georgia, United States

REFERENCES:
- [Background] Ji S, Long Q, Newport DJ, Na H, Knight B, Zach EB, Morris NJ, Kutner M, Stowe ZN. Validity of depression rating scales during pregnancy and the postpartum period: impact of trimester and parity. J Psychiatr Res. 2011 Feb;45(2):213-9. doi: 10.1016/j.jpsychires.2010.05.017. Epub 2010 Jun 9. PMID 20542520
- [Background] Miller AM, Hogue CJ, Knight BT, Stowe ZN, Newport DJ. Maternal expectations of postpartum social support: validation of the Postpartum Social Support Questionnaire during pregnancy. Arch Womens Ment Health. 2012 Aug;15(4):307-11. doi: 10.1007/s00737-012-0287-x. Epub 2012 May 16. PMID 22588510
- [Background] Newport DJ, Ji S, Long Q, Knight BT, Zach EB, Smith EN, Morris NJ, Stowe ZN. Maternal depression and anxiety differentially impact fetal exposures during pregnancy. J Clin Psychiatry. 2012 Feb;73(2):247-51. doi: 10.4088/JCP.10m06783. Epub 2011 Nov 29. PMID 22152400
- [Background] Schroeder JW, Conneely KN, Cubells JC, Kilaru V, Newport DJ, Knight BT, Stowe ZN, Brennan PA, Krushkal J, Tylavsky FA, Taylor RN, Adkins RM, Smith AK. Neonatal DNA methylation patterns associate with gestational age. Epigenetics. 2011 Dec;6(12):1498-504. doi: 10.4161/epi.6.12.18296. PMID 22139580
- [Background] Monk C, Newport DJ, Korotkin JH, Long Q, Knight B, Stowe ZN. Uterine blood flow in a psychiatric population: impact of maternal depression, anxiety, and psychotropic medication. Biol Psychiatry. 2012 Sep 15;72(6):483-90. doi: 10.1016/j.biopsych.2012.05.006. Epub 2012 Jun 12. PMID 22695184
- [Background] Schroeder JW, Smith AK, Brennan PA, Conneely KN, Kilaru V, Knight BT, Newport DJ, Cubells JF, Stowe ZN. DNA methylation in neonates born to women receiving psychiatric care. Epigenetics. 2012 Apr;7(4):409-14. doi: 10.4161/epi.19551. Epub 2012 Apr 1. PMID 22419064
- [Background] Lusby CM, Goodman SH, Bell MA, Newport DJ. Electroencephalogram patterns in infants of depressed mothers. Dev Psychobiol. 2014 Apr;56(3):459-73. doi: 10.1002/dev.21112. Epub 2013 Jul 12. PMID 23852456
- [Background] McConathy J, Capello C, Jarkas N, Stowe ZN, Owens MJ. Preparation of antidepressants for use in preclinical research. Int J Neuropsychopharmacol. 2007 Dec;10(6):759-63. doi: 10.1017/S1461145706007474. Epub 2007 Jan 4. PMID 17201995
- [Background] Capello CF, Bourke CH, Ritchie JC, Stowe ZN, Newport DJ, Nemeroff A, Owens MJ. Serotonin transporter occupancy in rats exposed to serotonin reuptake inhibitors in utero or via breast milk. J Pharmacol Exp Ther. 2011 Oct;339(1):275-85. doi: 10.1124/jpet.111.183855. Epub 2011 Jul 20. PMID 21775476
- [Background] Bourke CH, Capello CF, Rogers SM, Yu ML, Boss-Williams KA, Weiss JM, Stowe ZN, Owens MJ. Prenatal exposure to escitalopram and/or stress in rats: a prenatal stress model of maternal depression and its treatment. Psychopharmacology (Berl). 2013 Jul;228(2):231-41. doi: 10.1007/s00213-013-3030-z. Epub 2013 Feb 24. PMID 23436130
- [Background] Smith AK, Newport DJ, Ashe MP, Brennan PA, Laprairie JL, Calamaras M, Nemeroff CB, Ritchie JC, Cubells JF, Stowe ZN. Predictors of neonatal hypothalamic-pituitary-adrenal axis activity at delivery. Clin Endocrinol (Oxf). 2011 Jul;75(1):90-5. doi: 10.1111/j.1365-2265.2011.03998.x. PMID 21521269
- See also: Click here for the Women's Mental Health Program Web site — http://www.emorywomensprogram.org